CLINICAL TRIAL: NCT02379325
Title: 4-Weeks Intervention of Mobile Phone Text Messaging (Let's Quit!) on Smoking Cessation Among University Students: A Non Randomized Controlled Trial
Brief Title: Text Message Stop Smoking Among Young Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Lets Quit
Record Dates: First submitted 2015-02-05; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Young Adult Behavioral Change

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lets Quit (Experimental): Given text message
  Interventions: Behavioral: Lets Quit; Behavioral: pamphlets material
- Pamplets education (Active Comparator): Given pamplets on smoking and complication
  Interventions: Behavioral: Lets Quit; Behavioral: pamphlets material

INTERVENTIONS:
Behavioral: Lets Quit — Five tracks were created including "Not Ready", "Beginner", "Advance", "Relapse", and "Distraction". The "Distraction" track was combined with all of the other remaining 4 tracks. It was aimed as a distraction (as the name indicated) method to lighten the participants mood. It consisted of general information such as sports, fashion, dining, movies, and travelling.
Behavioral: pamphlets material — Given pamphlets material on smoking and complication

SUMMARY:
Smoking cessation is a priority for preventing smoking-attributable disease and reducing its burden. Quitting smoking at any age confers substantial and immediate health benefits, including reduced risks of stroke, cardiovascular disease and smoking-related cancers, and quitting smoking by the age of 30 reduces the risk of dying from tobacco-related diseases by almost 90%. The World Bank suggests that if adult cigarette consumption were to decrease by half in the year 2020, approximately 180 million tobacco-attributable deaths could be avoided. Therefore, promotion of smoking cessation has been proposed as a primary focus of tobacco control efforts, especially in developing countries where smoking prevalence and cigarette consumption are both still relatively high

DETAILED DESCRIPTION:
most risk factors are associated with more than one disease, and targeting those factors can reduce multiple causes of disease. Since smoking has 9% contributions on the leading global risk towards mortality in the world and this risk factor has resulted in multiple causes of disease for example, lung cancer, heart disease, stroke, chronic respiratory disease and other conditions therefore by quantifying the impact of this risk factors on diseases, may help to decrease the number of burden disease that is caused by smoking. University students age of 18 -24 are among the group of age that has the highest prevalence on smoking, thus it is necessary to targeting the high-risk people, who are most likely to benefit from the intervention. Population-based strategies seek to change the social norm by encouraging an increase in healthy behavior and a reduction in health risk. University students are in transition between the adolescence and early adulthood and developed unhealthy behaviors like cigarette smoking

ELIGIBILITY:
Inclusion Criteria:

* Smokers aged 18 - 24 years old
* Owned a mobile phone with text messaging capabilities
* Intention to quit
* No current use of nicotine replacement treatment or bupropion in the past month
* Not in treatment for any substance abuse disorder within the past year

Exclusion Criteria:

* Not a smoker
* No desire to quit smoking-
* Who unwillingly to participate in this study

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Quit rates | 2 months
Time-line follow-back (TLFB) | 2 months
The Fagerstrom Test for Nicotine Dependence | 2 months
CO level | 2 months